CLINICAL TRIAL: NCT03095378
Title: Evaluation of Root Coverage by Subepithelial Connective Graft Associated to Root Conditioning by Citric Acid Plus Tetracycline and Antimicrobial Photodynamic Therapy: A Randomized Clinical Trial
Brief Title: Evaluation of Root Coverage by Connective Graft and Different Root Conditioning Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BauruSchoolDentistryPDT
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Gingival Recession
Keywords: gingival recession
MeSH Terms: conditions — Gingival Recession | interventions — Citric Acid; Tetracycline

STUDY DESIGN:
Intervention Model Description: Interventions in different patients
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor did not have access to patient's records
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Root treatment with scaling and root planing.
  Interventions: Procedure: Control
- Citric acid plus tetracycline (Experimental): Root treatment with 50% citric acid plus 10% tetracycline, pH1, passive application for 90s.
  Interventions: Procedure: citric acid plus tetracycline
- Antimicrobial photodynamic therapy (Experimental): Antimicrobial photodynamic therapy with toluidine blue O (100ug/ml - 60s pre-irradiation - pH4) and red laser (660nm, 30 milliwatts, 45 joules per square centimeter, sweeping mode, 90s)
  Interventions: Procedure: antimicrobial photodynamic therapy

INTERVENTIONS:
Procedure: Control — Periodontal plastic surgery aiming root coverage by palatal connective tissue graft. Root treatment with scaling and root planing
  Arms: Control
Procedure: citric acid plus tetracycline — Periodontal plastic surgery aiming root coverage by palatal connective tissue graft. Root treatment with citric acid plus tetracycline
  Arms: Citric acid plus tetracycline
Procedure: antimicrobial photodynamic therapy — Periodontal plastic surgery aiming root coverage by palatal connective tissue graft. Root treatment with antimicrobial photodynamic therapy
  Arms: Antimicrobial photodynamic therapy

SUMMARY:
The aim of this study was to evaluate the effect of two root-conditioning agents used in conjunction with subepithelial connective graft technique on root coverage outcomes. One is citric acid plus tetracycline and the other is antimicrobial photodynamic therapy.

DETAILED DESCRIPTION:
Citric acid plus tetracycline has properties of root surface decontamination, surface demineralization and exposure of collagen fibers.

Antimicrobial photodynamic therapy has been widely used in Periodontics to obtain reduction of periodontopathogenic bacteria with absence of systemic side effects and minimal bacterial resistance. Also, it has properties of root demineralization and exposure of collagen fibers. These properties may enhance root coverage in procedures of subepithelial connective graft.

ELIGIBILITY:
Inclusion Criteria:

* Gingival recession - Miller's class I or II (2 to 5 mm of height) at least in one tooth
* Indication of root coverage by dentin hypersensitivity or esthetic

Exclusion Criteria:

* Smokers
* Pregnancy
* Systemic medication use that could impair wound healing or surgery procedure
* Systemic diseases as diabetes, uncontrolled hypertension, coagulation diseases, kidney diseases.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Total root coverage measured with a periodontal probe in mm | one year
  Distance from cemento-enamel junction to gingival margin = 0 mm

SECONDARY OUTCOMES:
Keratinized mucosa width measured with a periodontal probe in mm | one year
  Ideal if keratinized mucosa width > 5mm
Dentin hypersensitivity measured by applying an air jet on teeth and patient fills up a visual analogue scale | one year
  Ideal if scale = 0

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damante CA, Ducati P, Ferreira R, Salmeron S, Zangrando MSR, de Rezende MLR, Sant'Ana ACP, Greghi SLA, Magalhaes AC. In vitro evaluation of adhesion/proliferation of human gingival fibroblasts on demineralized root surfaces by toluidine blue O in antimicrobial photodynamic therapy. Photodiagnosis Photodyn Ther. 2016 Mar;13:303-307. doi: 10.1016/j.pdpdt.2015.08.009. Epub 2015 Sep 7. PMID 26358636
- [Background] Karam PS, Sant'Ana AC, de Rezende ML, Greghi SL, Damante CA, Zangrando MS. Root surface modifiers and subepithelial connective tissue graft for treatment of gingival recessions: a systematic review. J Periodontal Res. 2016 Apr;51(2):175-85. doi: 10.1111/jre.12296. Epub 2015 Jun 11. PMID 26095265